CLINICAL TRIAL: NCT04805697
Title: Fermented Grape Drinks Made of Fermented Grapes With Fruit and Vegetable Powder to Explore Whether it Can Improve the Skin's Condition and Achieve Anti-inflammatory Effects.
Brief Title: Fermented Grape Combined With Fruits and Vegetables Drink on Anti-aging and Anti-inflammatory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-054-B
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): subjects drank 50 ml , 1 bottle a day for 8 week
  Interventions: Dietary Supplement: placebo group
- fermented grape drinks (Experimental): subjects drank 50 ml , 1 bottle a day for 8 week
  Interventions: Dietary Supplement: fermented grape drinks

INTERVENTIONS:
Dietary Supplement: placebo group — subjects drank 50 ml , 1 bottle a day for 8 week
  Arms: placebo group
Dietary Supplement: fermented grape drinks — subjects drank 50 ml , 1 bottle a day for 8 week
  Arms: fermented grape drinks

SUMMARY:
60 subjects were recruited and divided into placebo group and fermented grape drinks group.

DETAILED DESCRIPTION:
In this study, using a fermented grape drinks made of fermented grapes with fruit and vegetable powder to explore whether it can improve the skin's condition and achieve anti-inflammatory effects. Sixty subjects were recruited and divided into placebo group and fermented grape drinks group. After drinking for 8 weeks, skin test and blood biochemical analysis were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Dry skin.
2. Rough skin
3. Large pores
4. Dark yellow complexion
5. Sagging skin

Exclusion Criteria:

1. Skin disorders
2. Liver diseases
3. Kidney diseases
4. Allergy to cosmetics, drugs, or foods
5. Pregnant and lactating women
6. People who had any cosmetic procedures before 4 weeks of the study
7. Area of facial spot over 3 cm2
8. Vegan
9. People who took collagen supplements in the past 3 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
skin brightness | 8 week
  The subjects divided into a placebo group (n=30) and an experimental group (n=30). Each subject was informed to consume one bottle of a 50 mL of grape drink or a placebo drink daily for 8 weeks, then using corneometer CM825 to examine skin brightness (The higher the value, the more water content, C.U., corneometer units )
skin elasticity | 8 week
  The subjects divided into a placebo group (n=30) and an experimental group (n=30). Each subject was informed to consume one bottle of a 50 mL of grape drink or a placebo drink daily for 8 weeks, then using cutometer dual MPA580 to examine skin elasticity (The closer the R2 value is to 1, the better the elasticity and no unit)
skin moisture | 8 week
  The subjects divided into a placebo group (n=30) and an experimental group (n=30). Each subject was informed to consume one bottle of a 50 mL of grape drink or a placebo drink daily for 8 weeks, then using probe system GL2000 & MPA10 to examine skin moisture (The higher the value, the higher the gloss, no unit)
skin spot | 8 week
  The subjects divided into a placebo group (n=30) and an experimental group (n=30). Each subject was informed to consume one bottle of a 50 mL of grape drink or a placebo drink daily for 8 weeks, then usig VISIA-CR to examine skin spot (The higher the value, the larger the pore area, mm2)
skin wrinkle | 8 week
  The subjects divided into a placebo group (n=30) and an experimental group (n=30). Each subject was informed to consume one bottle of a 50 mL of grape drink or a placebo drink daily for 8 weeks, then using VISIOSCAN-VC20 to examine skin wrinkle (The higher the value, the more wrinkles, surface evaluation of wrinkles, SEW)
inflammatory cytokines | 8 week
  The subjects divided into a placebo group (n=30) and an experimental group (n=30). Each subject was informed to consume one bottle of a 50 mL of grape drink or a placebo drink daily for 8 weeks, then using ELISA kit to examine inflammatory cytokines (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Ph.D, Study Director — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Research & Design Center, TCI CO., Ltd, Taipei, Taiwan